CLINICAL TRIAL: NCT04691765
Title: A Phase 1 Trial of Anakinra in Previously Untreated Chronic Lymphocytic Leukemia Patients at Risk for Progression
Brief Title: Anakinra in Previously Untreated Chronic Lymphocytic Leukemia Patients
Acronym: Anakinra
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. David Spaner (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor-Investigator, Dr. David Spaner, Haematologist, Senior Scientist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Anakinra
Record Dates: First submitted 2020-11-23; First posted 2020-12-31 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2020-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; Chronic Lymphocytic Leukemia; Anakinra; type 1 interferon; IFN; dose-limiting toxicity; Kineret
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: The trial will involve 12 patients in a standard dose escalation design. The first cohort of 4 patients will start at 100 mg SC daily, the dose approved for rheumatoid arthritis. If no dose limiting toxicities are experienced by these patients during the first cycle of treatment, then the next cohort of up to 4 patients will be treated at 100 mg SC twice daily (BID). The third cohort of up to 4 patients will be treated at 200 mg BID SC daily, to approximate doses used to treat inflammopathies such as Cryopyrin-Associated Periodic Syndromes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 100 mg SC (Experimental): 100 mg of Kineret (anakinra) will be administered sub-subcutaneously once a day for 28 days (1 cycle) with a maximum of 7 cycles (28 weeks of treatment)
  Interventions: Drug: Kineret
- 100 mg SC BID (Experimental): 100 mg of Kineret (anakinra) will be administered sub-subcutaneously twice a day for 28 days (1 cycle) with a maximum of 7 cycles (28 weeks of treatment)
  Interventions: Drug: Kineret
- 200 mg SC BID (Experimental): 200 mg of Kineret (anakinra) will be administered sub-subcutaneously twice a day for 28 days (1 cycle) with a maximum of 7 cycles (28 weeks of treatment)
  Interventions: Drug: Kineret

INTERVENTIONS:
Drug: Kineret — escalating doses of drug will be administered to 3 groups of 4 patients for 7 months
  Other Names: Anakinra

SUMMARY:
This is a phase I trial of the IL-1 receptor antagonist anakinra in chronic lymphocytic leukemia patients who are predicted to eventually require first-line therapy based on conventional clinical criteria. Three groups of 4 patients will be injected subcutaneously with either 100 mg daily or 100 mg twice daily or 200 mg twice daily for 7 cycles of 4 weeks each to determine the dose-limiting toxicity of anakinra in this population. Clinical responses will be determined by conventional IWCLL criteria. It is hoped anakinra will prevent disease progression with little toxicity. The study is anticipated to be completed within a year.

DETAILED DESCRIPTION:
To avoid unnecessary toxicity from treatments that do not cure, patients with chronic lymphocytic leukemia (CLL) patients are traditionally observed until they develop symptoms that justify first-line therapy. This period of observation is called "watch and wait". Treatment of symptomatic CLL has improved significantly with new drugs such as ibrutinib that provide disease control previously impossible with standard chemotherapy. Unfortunately, these drugs rarely cure and outcomes are poor once they stop working. There is a need for strategies to prevent disease progression during "watch and wait" in order to extend survival and improve the lives of CLL patients.

It has been found that CLL cells from many patients spontaneously make the cytokine interleukin-1 (IL-1). When IL-1 is blocked by the IL-1 receptor antagonist anakinra, CLL cells release high amounts of type 1 interferon (IFN). Since IFN produced at sufficient levels for appropriate times activates immune responses that may prevent progression of cancer and anakinra has a favorable toxicity profile, the hypothesis of this trial is that anakinra administered in the "watch and wait" period may clear CLL cells before they can cause symptoms.

The hypothesis will be addressed in a phase 1 clinical trial. The primary objective is to determine the dose-limiting toxicity (DLT) of anakinra, which has not been established previously in this patient population. The secondary objectives are to determine the effect on disease burden. Anakinra will be provided by Sobi and clinical trial costs supported by the Sunnybrook hematology site group. The trial will involve 3 cohorts of 4 patients in a standard phase 1 design. Eligible patients will be on "watch and wait" but expected to inevitably require treatment as predicted by unmutated IGHV status, presence of lymphadenopathy or splenomegaly, circulating CLL counts greater than 30x106 cells/ml, or IgG levels less than 8 g/L. Cohorts will be treated with 100 mg subcutaneously (SC BID) daily, the dose approved for rheumatoid arthritis, 100 mg SC BID, or 200 mg BID, to approximate doses for genetic inflammopathies. Anakinra will be given daily for seven 4-week cycles based on experience with other immunomodulatory drugs that suggest an average time to best response is ~7 months. Responses will be determined by conventional criteria based on decreases in circulating CLL cell numbers and radiologic measurements of lymphadenopathy. Anakinra will be considered ineffective if no clinical responses are observed after 7 cycles. Based on Gehan criteria, a new drug must show activity in at least 1/13 patients to justify further testing.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CLL meeting published diagnostic criteria: monoclonal B cells (either kappa or lambda light chain restricted) that are clonally co-expressing at least 1 B-cell marker (CD19 or CD20) and CD5 with prolymphocytes comprising no more than 55% of blood lymphocytes.
2. Unmutated IGHV status or Rai stage 2-4 or Rai stage 0-1 with blood lymphocytes greater than 30 x 106 cells/ml or IgG less than 8 g/L.
3. Not currently treated with other agents for CLL.
4. Serum bilirubin, and alanine transferase less than or equal to twice the upper limit of normal.
5. Platelets > or equal to 75x109/L. ANC > or equal to.75x109/L. Hemoglobin > or equal to 65 g/L
6. Age>18 years old
7. ECOG<2

Exclusion Criteria:

1. Patients with inadequate bone marrow reserve at baseline visit as demonstrated by at least one of the following: a. ANC<.75x109/L b. platelets <75x109/L without the assistance of growth factors, thrombopoietic factors, or platelet transfusions. C. hemoglobin <65 g/L despite transfusions.
2. Patients who have or have had progressive multifocal leukoencephalopathy (PML).
3. Patients with clinically significant bacterial, fungal, parasitic or viral infection, which require therapy. Patients with acute bacterial infections requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed.
4. Patients with known active hepatitis A, B, C or who are HIV-positive or who are at risk for HBV reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Prior test results obtained as part of standard of care that confirm a subject is immune and not at risk for reactivation (ie, hepatitis B surface antigen negative, surface antibody positive) may be used for purposes of eligibility and tests do not need to be repeated. Subjects with prior positive serology results must have negative polymerase chain reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.
5. Primary immunodeficiency such as X-linked agammaglobulinemia or common variable immunodeficiency.
6. Patients with active and inactive ('latent') tuberculosis infection or suspicion of active tuberculosis. If no suspicion of active tuberculosis, testing is not required.
7. Involvement of the central nervous system by lymphoma or leukemia.
8. Richter's transformation or prolymphocytic leukemia.
9. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
10. Use of glucocorticoids above the equivalent of 10 mg of prednisone daily within 4 weeks prior to treatment with anakinra. Patients cannot previously have taken drugs or antibodies normally used to treat CLL (eg. chlorambucil, fludarabine, cyclophosphamide, bendamustine, rituximab, ofatumumab, ibrutinib, venetoclax).
11. Major surgery within 4 weeks prior to treatment.
12. Patients with a history of malignancy in the past 3 years except for treated, early-stage squamous or basal cell carcinoma, carcinoma-in-situ of the cervix, or low-risk prostate cancer after curative therapy.
13. History or current diagnosis of uncontrolled or significant cardiac disease, including any of the following: a. myocardial infarction within last 6 months. b. uncontrolled congestive heart failure. c. unstable angina within last 6 months. d. exertional angina. e. clinically significant (symptomatic) cardiac arrhythmias (eg. bradyarrhythmias, sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemarker).
14. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
15. Presence of severe renal function impairment (estimated creatinine clearance <30 mL/min/1.73m2).
16. Patients with mild, moderate, or severe hepatic impairment or inadequate liver function defined by any of direct bilirubin, alanine amino transferase (ALT), or aspartate aminotransferase (AST)>2.5 x upper limit of normal (ULN). Patients with Child-Pugh score >5 are also excluded.
17. Patients under ongoing treatment with another investigational medication or having been treated with an investigational medication within 30 days of screening or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
18. Significant concurrent, uncontrolled medical condition which, in the investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.
19. Subjects who are unable to comprehend or are unwilling to sign an informed consent form (ICF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Safety and dose limiting toxicities of anakinra in CLL patients | 1 year
  The primary endpoints relate to safety and tolerability of anakinra in this patient, including numbers of patients with treatment-related adverse events (AEs) as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Efficacy of anakinra in CLL patients | 1 year
  Efficacy, defined as the proportion of patients with complete response (CR) or proportion of patients with partial response as defined by the NCI-WG guidelines on CLL.

CONTACTS AND LOCATIONS:
Overall Officials: David Spaner, MD, Principal Investigator — Sunnybrook Health Sciences Centre